CLINICAL TRIAL: NCT01359618
Title: A Single-centre, Randomised, Double-blind, Placebo Controlled Phase I Study in Two Parts: Part A to Assess a Safe and Tolerable Supratherapeutic Dose of TC-5214 After Single Ascending Oral Doses in Healthy Male Subjects, Followed by Part B: A Four-period Double-dummy Crossover Study to Investigate the Effect of 2 Single Doses (Therapeutic and Supratherapeutic) of TC-5214 on the QT/QTc Interval, Compared to Placebo, Using Moxifloxacin (Avelox®) as a Positive Control, in Healthy Male Subjects
Brief Title: Determining Highest Dose Administration of TC-5214 and Evaluating Effect on the Electrical Activity in the Heart
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to terminate
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D4130C00009
Record Dates: First submitted 2011-04-28; First posted 2011-05-25 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Healthy Male
Keywords: Phase I; Safety; tolerability; healthy; major depressive disorder; thorough QT; maximum tolerated dose; elimination; heart electrical signal
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A 1 (Experimental): TC-5214
  Interventions: Drug: TC-5214
- Part A 2 (Experimental): TC-5214 placebo
  Interventions: Other: Placebo comparator
- Part B 1 (Experimental): TC-5214 8 mg + moxifloxacin placebo
  Interventions: Drug: TC-5214; Other: Moxifloxacin placebo comparator
- Part B 2 (Experimental): TC-5214 supratherapeutic dose + moxifloxacin placebo
  Interventions: Drug: TC-5214; Other: Moxifloxacin placebo comparator
- Part B 3 (Active Comparator): TC-5214 placebo + moxifloxacin 400 mg
  Interventions: Other: Placebo comparator; Drug: Moxifloxacin
- Part B 4 (Placebo Comparator): TC-5214 placebo + moxifloxacin placebo
  Interventions: Other: Placebo comparator; Other: Moxifloxacin placebo comparator

INTERVENTIONS:
Drug: TC-5214 — Single dose, oral tablets
  Arms: Part A 1; Part B 1; Part B 2
Other: Placebo comparator — Single dose, oral tablets
  Arms: Part A 2; Part B 3; Part B 4
Drug: Moxifloxacin — Single dose, oral encapsulated tablet
  Other Names: Avelox®
  Arms: Part B 3
Other: Moxifloxacin placebo comparator — Single dose, oral encapsulated tablet
  Arms: Part B 1; Part B 2; Part B 4

SUMMARY:
This is a two part study. Part A will determine the maximum tolerated dose of TC-5214 administered to healthy male subjects in single ascending oral doses. This part of the study will define the highest dose of TC-5214 to be administered in Part B. Part B of this study will investigate the effect of TC-5214 on the electrical activity of the heart following single oral administration. The study will be carried out healthy male subjects in a four period crossover study with TC-5214 compared to placebo and oral moxifloxacin as a positive control. The safety, tolerability and pharmacokinetics of TC-5214 will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male 18 to 50 years old inclusive with suitable veins for cannulation or repeated venipuncture
* Have a body mass index (BMI) between 19 and 30 kg/m2 inclusive and weigh at least 50 kg
* Male subjects should be willing to use a double barrier method of contraception (condom with spermicide) from the first dose of investigational product until 3 months after the last dose of investigational product
* Be able to understand and comply with the requirements of the study as judged by the investigator

Exclusion Criteria:

* History of any clinically significant medical, neurologic or psychiatric disease or disorder which, in the opinion of the Investigator and Sponsor may either put the subject at risk because of participation in the study, or influence the results of the subject's ability to participate in the study
* History or presence of gastrointestinal (including irritable bowel disease), hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of study drug. Subjects with a history of surgery on the gastrointestinal tract (not including appendectomy or cholecystectomy) should also be excluded
* History of seizure activity, including febrile seizures
* Prolonged QTcF >450 ms or shortened QTcF <340 ms, or family history of Long QT Syndrome
* Use of concomitant medications that prolong QT/QTc interval

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Part A: To examine the safety and tolerability of TC-5214. The following assessments will be measured and reported: The number of participants with adverse events | Up to 24 hours
Part A: To examine the safety and tolerability of TC-5214. The following assessments will be measured and reported: A change from baseline in laboratory assessments. | Up to 24 hours
Part A: To examine the safety and tolerability of TC-5214. The following assessments will be measured and reported: A change from baseline in vital signs. | Up to 24 hours
Part A: To examine the safety and tolerability of TC-5214. The following assessments will be measured and reported: A change from baseline in electrocardiogram (ECG). | Up to 24 hours
Part A: To examine the safety and tolerability of TC-5214. The following assessments will be measured and reported: A change from baseline in physical examination. | Up to 24 hours
Part B: The maximum mean change in time-matched ECG interval, measured from the onset of the QRS complex to the T point, using the best heart rate correction method (QTc). | Up to 24 hours

SECONDARY OUTCOMES:
Part A: TC-5214 Plasma and urine pharmacokinetic variable to be measured: including, C max, time to C max, Area Under Curve (AUC) (0-t), terminal half life, cumulative amount of drug excreted unchanged into urine from zero to time and renal clearance | Up to 72 Hours
Part B: A change in the maximum of the mean change in time-matched ECG interval, measured from the onset of the QRS complex | Up to 24 Hours
Part B: Assay sensitivity by measuring the effect of moxifloxacin 400 mg on QTc compared to placebo | Up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hans A Eriksson, MD, PhD, MBA, Study Director — AstraZeneca; Darren Wilbraham, MBBS DCPSA, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital; Brendan Smyth, MD, Study Chair — AstraZeneca
Locations (1):
- Research Site, London, United Kingdom